CLINICAL TRIAL: NCT03218358
Title: Effect of the Intra-abdominal Pressure on the Risk of Delirium in Mechanically Ventilated Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, Principal investigator, Assiut University
Other Study IDs: delirium & IAP
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Delirium; Intraabdominal Hypertension; Mechanical Ventilation Complication
MeSH Terms: conditions — Delirium; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
intra-abdominal hypertension (IAH) and delirium are serious, high-frequency complications in intensive care unit (ICU) patients. The consequences of the complication range from high morbidity and mortality to a greater need for nursing care. We hypothesize that there could be a correlation between IAH and incidence of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders on mechanical ventilation

Exclusion Criteria:

* age under 18 years, use of muscle relaxants, abdominal operation within the previous 3 months, acute peritonitis, and abdominal mass, acute injury to the urinary bladder, acute cystitis, neurogenic bladder, pelvic hematoma, and pelvic fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 critically ill patients that remained more than 48 hours at trauma and general ICU without apparent risk factors for IAH other than the use of MV
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
delirium | 3 days
  NEECHAM confusion scale will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No